CLINICAL TRIAL: NCT04111653
Title: Exploration of the Transfer of Barium From Thermal Mud (T2BT Study)
Brief Title: Exploration of the Transfer of Barium From Thermal Mud
Acronym: T2BT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association Francaise pour la Recherche Thermale (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019-A01614-53
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Mud Therapy
Keywords: mud therapy; natural mineral water; barium; poultices; skin transfer
MeSH Terms: interventions — Mud Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): Healthy volunteers
  Interventions: Other: Mud therapy

INTERVENTIONS:
Other: Mud therapy — Application of sludge poultice

SUMMARY:
It involves conducting a clinical study on a population of healthy volunteers (age between 18 and 30 years) without direct benefit for the subject to explore a transfer of barium in the blood and urine following applications of thermal mud. The main objective is to highlight an increase in serum barium level of at least twice.

DETAILED DESCRIPTION:
The presence of barium in thermal clays was noted by the ARS (french administration) who interviewed the Directorate General of Health (DGS); the latter seized the National Academy of Medicine (June 2016) which reported in February 2017.

In this report it was stated that there was no argument in favor of toxic phenomena related to the presence of barium but that it was appropriate, in particular, to evaluate a possible passage of barium in the skin in subjects who are treated with thermal mud

* by observing, where appropriate, an increase in serum and urinary barium levels in the subjects concerned and
* by measuring a possible depletion of barium in the sludge used. The DGS validated the various recommendations of the Academy and asked, in January 2018, the National Council of Thermal Establishments (CNETH) to implement the recommendations of the Academy.

It will therefore be a prospective before-after interventional study, implementing 15 daily applications of 6 mud poultices made with a clay used as thermal clay and containing appreciable barium levels.

A surveillance will be put in place with the event of suspected event, the volunteer can then be seen by a doctor.

ELIGIBILITY:
Inclusion Criteria:

* volunteers, healthy (without known and / or treated disease)
* 18 to 30 years old,
* men and women, who can give their informed consent, presenting the elements of cutaneous and general tolerance of sludge applications
* patient affiliated to a social security scheme

Exclusion Criteria:

* subject who can not give informed consent
* pregnant woman ; woman of childbearing years not wishing to have contraception available for the duration of the trial
* subject to a legal protection measure or a judicial review, subject having a known allergy to a heavy metal, a BMI greater than 30
* a characterized contact eczema, an active dermatosis, an acute affection, a disorder of the cutaneous sensitivity, an intolerance to the heat
* heart, kidney or lung disease that may be decompensated with the use of hot products
* a progressive disease (inflammatory, infectious or tumoral) potentially liable to worsen with the application of thermal physical agents

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of the plasma level of barium | 3 weeks
  Plasma level of barium

SECONDARY OUTCOMES:
Measurement of the urinary rate of barium | 3 weeks
  Urinary rate of barium
Plasma level of barium exceeds the level deemed tolerable by INRS (French Institute for Research and Security) | 3 weeks
  plasma levels of barium
Number of patients who doubles the urinary and plasma level of barium | 3 weeks
  plasma and urinary levels of barium

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Bauduer, Pr, Principal Investigator — Institut du thermalisme
Locations (1):
- Institut du Thermalisme, Dax, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roques CF, Trèves R, Queneau P, Bontoux D. Avis de l'académie nationale de médecine relatif à l'évaluation des risques sanitaires liés à la présence de baryum dans des argiles constitutives des boues thermales et à l'absence de contrôle sanitaire des boues thermales. Bull Acad Ntle Méd., , 201: 13-38, 2017.
- [Background] Ainouche R, Tabone W, Bouvier CE, Renaud V. Usage thérapeutique (des boues thermales), panorama du thermalisme français en 2013. Bulletin de l'AFTH (Association Française des Techniques Hydrothermales), 2014, n° 25, Symposium Utilisation des boues en établissement thermal, Enghien les Bains, Novembre 2013, pp. 7-11
- [Background] Gomes C, Carretero MI, Pozo M, Maraver F, Cantista P et al. Peloids and pelotherapy : historical evolution, classification and glossary. Applied clay science 75-76:28-38, 2013.
- [Background] Liu H, Zeng C, Gao SG, Yang T, Luo W, Li YS, Xiong YL, Sun JP, Lei GH. The effect of mud therapy on pain relief in patients with knee osteoarthritis: a meta-analysis of randomized controlled trials. J Int Med Res. 2013 Oct;41(5):1418-25. doi: 10.1177/0300060513488509. Epub 2013 Sep 5. PMID 24008567
- [Background] Roques CF. Mud Therapy. Data of clinical evidence. Balnea 10:57-62, 2015.
- [Background] Xiang J, Wu D, Li J. Clinical Efficacy of Mudpack Therapy in Treating Knee Osteoarthritis: A Meta-Analysis of Randomized Controlled Studies. Am J Phys Med Rehabil. 2016 Feb;95(2):121-31. doi: 10.1097/PHM.0000000000000354. PMID 26203645
- [Background] Roques CF, Queneau P. [SPA therapy for pain of patients with chronic low back pain, knee osteo-arthritis and fibromyalgia]. Bull Acad Natl Med. 2016 Mar;200(3):575-86; discussion 586-7. French. PMID 28644605
- [Background] World Health Organization (WHO) - 2001 - IPCS (International Programme on Chemical Safety) - Concise international chemical assessment document 33 - barium and barium compounds. 57 pp
- [Background] Conseil canadien des Ministres de l'environnement - Recommandations canadiennes pour la qualité des sols - environnement et santé humaine. Le baryum. Feuillet d'information 2013, 1 doc 11 pp
- [Background] Kravchenko J, Darrah TH, Miller RK, Lyerly HK, Vengosh A. A review of the health impacts of barium from natural and anthropogenic exposure. Environ Geochem Health. 2014 Aug;36(4):797-814. doi: 10.1007/s10653-014-9622-7. Epub 2014 May 21. PMID 24844320
- [Background] INRS - base de données de fiches toxicologiques. Baryum et composés. Fiche toxicologique complète n°125. 1 doc 12 pp, 2012
- [Background] Ding C, Pan Y, Zhang A, Zhu C, Liu D, Xu G, Zheng Y, Yan H. [Distribution of rubidium, cesium, beryllium, strontium, and barium in blood and urine in general Chinese population]. Zhonghua Lao Dong Wei Sheng Zhi Ye Bing Za Zhi. 2015 Dec;33(12):894-9. doi: 10.3760/cma.j.issn.1001-9391.2015.12.004. Chinese. PMID 27122328